CLINICAL TRIAL: NCT03816683
Title: Treatment Patterns, Outcomes, and Patient-Reported Health-Related Quality of Life: A Prospective Disease Registry of Patients With Mantle Cell Lymphoma Treated With Novel Agents
Brief Title: A Disease Registry of Patients With Mantle Cell Lymphoma
Acronym: SUMMIT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00004
Record Dates: First submitted 2018-12-10; First posted 2019-01-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Registry; MCL novel therapy; MCL treatment patterns; MCL reported outcomes
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort (registry) of MCL patients: Patients diagnosed with MCL who have initiated a novel therapy meeting inclusion/exclusion criteria in the past 6 months and treatment is ongoing at the time of enrollment.

SUMMARY:
The purpose of this study is to create a patient registry in order to assess treatment patterns, physician reported clinical outcomes and patient-reported health-related quality of life among patients diagnosed with Mantle Cell Lymphoma (MCL) who newly initiated a novel therapy in the past 6 months and whose treatment is ongoing at the time of enrollment.

DETAILED DESCRIPTION:
Newer targeted therapies (monotherapy or in combination with other agents) have been recently approved in the United States for the treatment of adult patients with mantle cell lymphoma (MCL) who have received at least 1 prior therapy. The approval of these newer therapies will have an impact on the treatment patterns, toxicity patterns, and outcomes in the MCL population. A prospective, observational study will help to better understand the evolving real-world treatment outcomes (including treatment patterns, reasons for discontinuation/dose reduction, treatment interruption or treatment switches), physician-reported clinical outcomes, and patient-reported symptoms and health-related quality of life (HRQoL) among patients diagnosed with Mantle Cell Lymphoma (MCL) who newly initiated a novel therapy in the past 6 months and whose treatment is ongoing at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Mantle Cell Lymphoma (MCL)
* Informed consent for participation
* Age ≥ 18 years old, as of the first observed diagnosis of MCL
* Patients for whom a clinical decision has been made to initiate novel therapy in the last 6 months, limited to the following novel agent categories:

  * Bcl-2 inhibitors
  * BTK inhibitors
  * Immunomodulatory agents
  * Phosphoinositide 3-kinase inhibitors The novel agent must have been granted approval in at least one haematological cancer. Treatment must be ongoing at the time of enrollment.

Exclusion Criteria:

• Patient is participating in a clinical study that prohibits participation in non-interventional studies, or where treatment is blinded, at the time of consent.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of MCL who have received any line of novel MCL treatment within the past 6 months (and treatment is ongoing at the time of enrollment).
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
The frequency and proportion of patients exposed to each novel agent therapy | 24 to 60 months
  MCL novel agent treatment types are part of the primary study objective relating to treatment patterns and will be descriptive only and use aggregated patient data.
The frequency and proportion of patients exposed to novel agent by therapy regimen | 24 to 60 months
  MCL treatment regimens are part of the primary study objective relating to treatment patterns and will be descriptive only and use aggregated patient data.
The frequency and proportion of patients exposed to novel agent by line of therapy | 24 to 60 months
  MCL treatment line is part of the primary study objective relating to treatment patterns and will be descriptive only and use aggregated patient data.
The frequency and proportion of patients exposed to novel agent by therapy class | 24 to 60 months.
  MCL treatment class is part of the primary study objective relating to treatment patterns and will be descriptive only and use aggregated patient data.
The rate of patients who change novel agent therapy dose (in months) | 24 to 60 months.
  Summarizing MCL novel agent treatment dose changes are part of the primary study objective relating to treatment patterns and will be descriptive only. Time-to-dose change will be assessed. The rate of dose modification (in months) will be estimated using aggregated patient data. Summary statistics (mean, SD, median, IQR, minimum, and maximum) will be used to describe time on a particular dose, which will be measured from the start of treatment until the date of dose change or death.
The rate of patients who interrupt novel agent therapy (in months) | 24 to 60 months
  Summarizing MCL treatment interruptions are part of the primary study objective relating to treatment patterns and will be descriptive only. The rate of treatment interruption (in months) will be estimated using aggregated patient data. Summary statistics (mean, SD, median, IQR, minimum, and maximum) will be used to describe time on therapy, which will be measured from the start of treatment until the date of interruption or death.
The rate of patients who discontinue novel agent therapy (in months) | 24 to 60 months
  Summarizing MCL treatment discontinuations are part of the primary study objective relating to treatment patterns and will be descriptive only. The rate of treatment discontinuation (in months) will be estimated using aggregated patient data. Reasons for discontinuations will be collected and summarized categorically. Summary statistics (mean, SD, median, IQR, minimum, and maximum) will be used to describe time on therapy, which will be measured from the start of treatment until the date of discontinuation or death.
The duration of MCL treatment | 24 to 60 months
  Summarizing MCL treatment duration is part of the primary study objective relating to treatment patterns and will be descriptive only. The duration and number of cycles of each targeted treatment (mean, SD, median, IQR, minimum, and maximum) will be summarized. Summary statistics (mean, SD, median, IQR, minimum, and maximum) will be used to describe time on therapy (in months), which will be measured from the start of treatment until the date of discontinuation, interruption, switch or death.
Estimate the overall response rate (ORR) among patients diagnosed with MCL and initiating treatment with novel therapies | 24 to 60 months.
  ORR will be measured as the frequency and proportion of patients with a complete or partial response based on physician assessment during the observation period.
Estimate the complete response rate (CR) among patients diagnosed with MCL and initiating treatment with novel therapies. | 24 to 60 months.
  The CR will be calculated as the frequency and proportion of patients with a complete response based on physician assessment during the observation period.
Estimate progression-free survival (PFS) among patients diagnosed with MCL and initiating treatment with novel therapies. | 24 to 60 months
  All survival outcome measures will be descriptive only. PFS will be calculated as the time from the start of novel MCL treatment until progression or death. Summary statistics (mean, median, SD, IQR, minimum and maximum) will be used to describe PFS. Kaplan-Meier curves will be used to graphically show PFS.
Estimate event-free survival (EFS) among patients diagnosed with MCL and initiating treatment with novel therapies. | 24 to 60 months
  All survival outcome measures will be descriptive only. EFS will be calculated as the time from the start of novel MCL treatment to disease progression, death, or discontinuation of treatment for any reason (eg, toxicity, patient preference, or initiation of a new treatment without documented progression).
Estimate overall survival (OS) among patients diagnosed with MCL and initiating treatment with novel therapies. | 24 to 60 months
  All survival outcome measures will be descriptive only. OS will be captured using summary statistics (mean, SD, median, IQR, minimum and maximum), which will be used to describe time from diagnosis to death, time from enrollment to death, time from index novel MCL treatment to death and time from second treatment (if applicable) to death. Kaplan-Meier curves will be used to graphically show patient survival.

SECONDARY OUTCOMES:
The frequency of adverse events (AEs) in patients with MCL, where the term AE is used to include both serious and non-serious AEs. | 24 to 60 months
  The frequency of patients with AEs will be tabulated from the start of index novel MCL treatment. AEs (both in terms of the MedDRA Preferred Terms (PTs) and Common Terminology Criteria for Adverse Events [CTCAE] grade) will be listed individually by patient and described by System Organ Class (SOC) and PT.
The proportion of adverse events (AEs) in patients with MCL, where the term AE is used to include both serious and non-serious AEs. | 24 to 60 months
  The proportion of patients with AEs will be calculated from the start of index novel MCL treatment. AEs (both in terms of the MedDRA Preferred Terms (PTs) and Common Terminology Criteria for Adverse Events [CTCAE] grade) will be listed individually by patient and described by System Organ Class (SOC) and PT.
Estimate the frequency of serious adverse events (SAEs) in patients with MCL | 24 to 60 months
  The proportion and frequency patients with SAEs will be tabulated from the start of index novel MCL treatment.
Estimate the frequency of reported serious adverse safety events and adverse events leading to treatment changes associated with novel agents in patients with MCL | 24 to 60 months
  The proportion and frequency of all SAEs and any AEs leading to treatment changes will be tabulated overall, and will also include the frequency and proportion of: (1) drug discontinuations, (2) dose interruptions or (3) dose changes.
Estimate the frequency and proportion of patients experiencing a clinical event of interest (related to MCL or MCL treatment) | 24 to 60 months
  The clinical events of interest that have an economic impact will be tabulated with the frequency and proportion of patients experiencing the event. Medical interventions used for managing clinical events of interest including but not limited to: diagnostic tests, procedures and medications.
Estimate the frequency and proportion of patients experiencing healthcare resource utilization (HCRU), such as inpatient or emergency department visits | 24 to 60 months
  Each type of physician visit will be tabulated at the aggregate level using the mean, SD, median, IQR, minimum and maximum. The total number of visits across all facilities will also be calculated.
Tabulate HRQoL responses for the validated EORTC QLC-C30 Patient Reported Outcome (PRO) in patients with MCL | 24 to 60 months
  Descriptive statistics for each validated PRO will include continuous measures (mean, median, SD, IQR, minimum, and maximum) or achievement of a particular threshold (frequency and proportion), if applicable. This study will collect patient perceptions of HRQoL based on PRO measures in patients with MCL by collecting the European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) on a quarterly basis. The EORTC QLQ-C30 has a recall/observation period during the past week. The questionnaire uses a 4-point Likert scale ranging from 1: "Not at all" to 4: "Very much," and scores by dimension range from 0 to 100.
Tabulate HRQoL responses for the three selected, validated PRO-CTCAE PRO measures in patients with MCL | 24 to 60 months
  Descriptive statistics for each validated PRO will include continuous measures (mean, median, SD, IQR, minimum, and maximum) or achievement of a particular threshold (frequency and proportion), if applicable. This study will collect patient perceptions of HRQoL by collecting the PRO version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) (3 questions regarding muscle pain, joint pain, heart palpitations) on a quarterly basis. The PRO-CTCAE is intended for individuals 18 years or older and has a recall of the past 7 days. Responses to each question are scored from 0 to 4 (in order of increasing frequency and severity).
Tabulate HRQoL responses for the validated PRO EuroQoL 5-Dimension 5-Level (EQ-5D-5L) in patients with MCL | 24 to 60 months
  Descriptive statistics for each validated PRO will include continuous measures (mean, median, SD, IQR, minimum, and maximum) or achievement of a particular threshold (frequency and proportion), if applicable. This study will collect patient perceptions of HRQoL based on PRO measures in patients with MCL by collecting the EQ-5D-5L on a quarterly basis. This questionnaire is comprised of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and 1 visual analog scale used to assess a patient's self-rated health. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A unique health state is defined by combining 1 level from each of the 5 dimensions. Each health state is referred to in terms of a 5-digit code.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hermann, Study Director — Senior Medical Director, Haematology
Locations (29):
- United States (29):
  - Research Site, Montgomery, Alabama
  - Research Site, Clovis, California
  - Research Site, Boulder, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Ann Arbor, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, East Syracuse, New York
  - Research Site, New York, New York
  - Research Site, Eugene, Oregon
  - Research Site, Danville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Ahn IE, Farooqui MZH, Tian X, Valdez J, Sun C, Soto S, Lotter J, Housel S, Stetler-Stevenson M, Yuan CM, Maric I, Calvo KR, Nierman P, Hughes TE, Saba NS, Marti GE, Pittaluga S, Herman SEM, Niemann CU, Pedersen LB, Geisler CH, Childs R, Aue G, Wiestner A. Depth and durability of response to ibrutinib in CLL: 5-year follow-up of a phase 2 study. Blood. 2018 May 24;131(21):2357-2366. doi: 10.1182/blood-2017-12-820910. Epub 2018 Feb 26. PMID 29483101
- [Background] AstraZeneca Pharmaceuticals LP. CALQUENCE® (acalabrutinib) prescribing information. October 2017.
- [Background] Chen Y, Wang M, Romaguera J. Current regimens and novel agents for mantle cell lymphoma. Br J Haematol. 2014 Oct;167(1):3-18. doi: 10.1111/bjh.13000. Epub 2014 Jun 28. PMID 24974852
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] ClinicalTrials.gov. Identifier NCT02756247. A Clinical Trial of Buparlisib and Ibrutinib in Lymphoma. Accessed 24 January 2018. Available from: https://clinicaltrials.gov/ct2/show/NCT02756247].
- [Background] ClinicalTrials.gov. Identifier NCT03112174. Study of Ibrutinib Combined with Venetoclax in Subjects with Mantle Cell Lymphoma (SYMPATICO). Accessed 24 January 2018. Available from: https://clinicaltrials.gov/ct2/show/NCT03112174.
- [Background] Collett D. Modelling Survival Data in Medical Research. 3rd edition. Boca Raton, FL: CRC press; 2015.
- [Background] de Claro RA, McGinn KM, Verdun N, Lee SL, Chiu HJ, Saber H, Brower ME, Chang CJ, Pfuma E, Habtemariam B, Bullock J, Wang Y, Nie L, Chen XH, Lu DR, Al-Hakim A, Kane RC, Kaminskas E, Justice R, Farrell AT, Pazdur R. FDA Approval: Ibrutinib for Patients with Previously Treated Mantle Cell Lymphoma and Previously Treated Chronic Lymphocytic Leukemia. Clin Cancer Res. 2015 Aug 15;21(16):3586-90. doi: 10.1158/1078-0432.CCR-14-2225. PMID 26275952
- [Background] EORTC Quality of Life Group. EORTC QLQ-C30 Version 3.0. 1995. Accessed 25 January 2018. Available from: http://groups.eortc.be/qol/eortc-qlq-c30.
- [Background] EuroQol Research Foundation. EQ-5D-5L: About. Version 18 April 2017. Accessed 25 January 2018. Available from: https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/.
- [Background] Martin P, Byrtek M, Dawson K, Ziemiecki R, Friedberg JW, Cerhan JR, Flowers CR, Link BK. Patterns of delivery of chemoimmunotherapy to patients with follicular lymphoma in the United States: results of the National LymphoCare Study. Cancer. 2013 Dec 1;119(23):4129-36. doi: 10.1002/cncr.28350. Epub 2013 Sep 4. PMID 24006156
- [Background] Mato AR, Nabhan C, Thompson MC, Lamanna N, Brander DM, Hill B, Howlett C, Skarbnik A, Cheson BD, Zent C, Pu J, Kiselev P, Goy A, Claxton D, Isaac K, Kennard KH, Timlin C, Landsburg D, Winter A, Nasta SD, Bachow SH, Schuster SJ, Dorsey C, Svoboda J, Barr P, Ujjani CS. Toxicities and outcomes of 616 ibrutinib-treated patients in the United States: a real-world analysis. Haematologica. 2018 May;103(5):874-879. doi: 10.3324/haematol.2017.182907. Epub 2018 Feb 1. PMID 29419429
- [Background] National Cancer Institute. Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) (version 1.0). Last updated 24 February 2017. Accessed 25 January 2018. Available from: https://healthcaredelivery.cancer.gov/pro- ctcae/overview.html.
- [Background] National Comprehensive Cancer Network (NCCN). NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) Non-Hodgkin's Lymphomas. 2014. Version 4.2014.
- [Background] Steiner RE, Romaguera J, Wang M. Current trials for frontline therapy of mantle cell lymphoma. J Hematol Oncol. 2018 Jan 27;11(1):13. doi: 10.1186/s13045-018-0556-x. PMID 29374487
- [Background] Tam CS, Roberts AW, Anderson M, Dawson S, Hicks R, Burbury K, et al. Combination ibrutinib (Ibr) and venetoclax (Ven) for the treatment of mantle cell lymphoma (MCL): primary endpoint assessment of the phase 2 AIM study. Hematol Oncol. 2017;35(S2):144-5.
- [Background] Teras LR, DeSantis CE, Cerhan JR, Morton LM, Jemal A, Flowers CR. 2016 US lymphoid malignancy statistics by World Health Organization subtypes. CA Cancer J Clin. 2016 Nov 12;66(6):443-459. doi: 10.3322/caac.21357. Epub 2016 Sep 12. PMID 27618563
- [Background] Wang M, Rule S, Zinzani PL, Goy A, Casasnovas O, Smith SD, Damaj G, Doorduijn J, Lamy T, Morschhauser F, Panizo C, Shah B, Davies A, Eek R, Dupuis J, Jacobsen E, Kater AP, Le Gouill S, Oberic L, Robak T, Covey T, Dua R, Hamdy A, Huang X, Izumi R, Patel P, Rothbaum W, Slatter JG, Jurczak W. Acalabrutinib in relapsed or refractory mantle cell lymphoma (ACE-LY-004): a single-arm, multicentre, phase 2 trial. Lancet. 2018 Feb 17;391(10121):659-667. doi: 10.1016/S0140-6736(17)33108-2. Epub 2017 Dec 11. PMID 29241979
- [Background] Witzig TE. Current treatment approaches for mantle-cell lymphoma. J Clin Oncol. 2005 Sep 10;23(26):6409-14. doi: 10.1200/JCO.2005.55.017. PMID 16155027
- [Background] Wu J, Liu C, Tsui ST, Liu D. Second-generation inhibitors of Bruton tyrosine kinase. J Hematol Oncol. 2016 Sep 2;9(1):80. doi: 10.1186/s13045-016-0313-y. PMID 27590878
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Younes A, Hilden P, Coiffier B, Hagenbeek A, Salles G, Wilson W, Seymour JF, Kelly K, Gribben J, Pfreunschuh M, Morschhauser F, Schoder H, Zelenetz AD, Rademaker J, Advani R, Valente N, Fortpied C, Witzig TE, Sehn LH, Engert A, Fisher RI, Zinzani PL, Federico M, Hutchings M, Bollard C, Trneny M, Elsayed YA, Tobinai K, Abramson JS, Fowler N, Goy A, Smith M, Ansell S, Kuruvilla J, Dreyling M, Thieblemont C, Little RF, Aurer I, Van Oers MHJ, Takeshita K, Gopal A, Rule S, de Vos S, Kloos I, Kaminski MS, Meignan M, Schwartz LH, Leonard JP, Schuster SJ, Seshan VE. International Working Group consensus response evaluation criteria in lymphoma (RECIL 2017). Ann Oncol. 2017 Jul 1;28(7):1436-1447. doi: 10.1093/annonc/mdx097. PMID 28379322
- [Background] Yun S, Vincelette ND, Acharya U, Abraham I. Risk of Atrial Fibrillation and Bleeding Diathesis Associated With Ibrutinib Treatment: A Systematic Review and Pooled Analysis of Four Randomized Controlled Trials. Clin Lymphoma Myeloma Leuk. 2017 Jan;17(1):31-37.e13. doi: 10.1016/j.clml.2016.09.010. Epub 2016 Sep 19. PMID 27780690
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220R00004&attachmentIdentifier=732f4282-643d-49e9-9437-315fbb0d03f3&fileName=AZMCL_CSR_V1.0_Final_30Sep2025_SYNOPSIS_ONLY.pdf&versionIdentifier=